CLINICAL TRIAL: NCT04631458
Title: A Study Assessing Morbidity and Portal Circulation in Patients With Myeloproliferative Neoplasms and Splanchnic Vein Thrombosis
Brief Title: Outcomes in Patients With Myeloproliferative Neoplasm and Splanchnic Vein Thrombosis
Acronym: Mascot
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: MPN-SVT v11; 02/Dec/2013
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Myeloproliferative Neoplasm; Splanchnic Vein Thrombosis; Splanchnic Venous Thrombosis; Myeloproliferative Disorders
Keywords: thrombosis; splanchnic; anticoagulation; TIPSS; myeloproliferative
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard of care. — Observational trial.

SUMMARY:
Patients with Myeloproliferative neoplasms are at particular risk for developing arterial and venous thrombosis, especially thrombosis in the splanchnic venous system. The patho-physiology and natural history of MPN related SVT is poorly understood and treatment algorithms vary greatly. This is of considerable importance since the morbidity and mortality in this group of patients is high. This study aims to observe patients with MPN related SVT over a period of five years to document their clinical progress. Methods of observation include clinical assessment, standard investigations and laboratory based research investigations

DETAILED DESCRIPTION:
Study Title Morbidity and portal circulation in patients with Myeloproliferative neoplasms and splanchnic vein thrombosis: Mascot Protocol No. MPN-SVT v11; 02/Dec/2013 Study Design Prospective observational longitudinal study of patients with MPN related splanchnic vein thrombosis(study group) and patients with MPN without SVT (control group) Study Participants Patients with myeloproliferative neoplasms (MPN) and splanchnic vein thrombosis (SVT), patients with MPN and splenomegaly.

Number of subjects 40 patients Follow-up duration 5 years Study duration January 2014- January 2019. Primary Objectives 1. To describe morbidity/portal circulation in the patient group over the 18m from baseline 2. To examine if there are changes in endpoints from baseline to 18m 3. To compare patients with MPN related SVT and MPN without SVT Secondary Objectives 1. To describe morbidity/portal circulation in the patient group over 5 years from baseline 2. To examine if there are changes in endpoints from baseline to 5 years 3. To assess the impact of treatment including cytoreductive therapy, Janus kinase (JAK) inhibition and antithrombotic treatment on end points.

4. To assess adequacy of anti-thrombotic agents with reference to recurrence, recanalisation and extension of splanchnic thrombosis, non-splanchnic thrombotic events and bleeding frequency.

Exploratory objectives 1. Assess the utility of endothelial colony assay as marker of disease 2. Assess the utility of adhesion molecules as markers of disease

Primary Endpoint Composite end point comprising occurrence or change in morbidity or portal circulation over 18 months Secondary Endpoint Occurence or change in morbidity or portal circulation over 3-5 years

ELIGIBILITY:
Inclusion Criteria:

1. MPN with SVT between 3 weeks to 5 years of diagnosis of SVT: study arm
2. MPN with palpable splenomegaly or enlarged by Ultrasound: control arm

Exclusion Criteria:

Age <18 years Patients with SVT without MPN

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: as above
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-11-12 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite end point comprising occurrence or change in morbidity or portal circulation over 18 months | 12-18 months from baseline
  analysed by radiologic investigations and clinical progress

SECONDARY OUTCOMES:
1. Occurrence or changes in morbidity over 5 years 2. Occurrence or changes in portal circulation over 5 years | 5 years from baseline
  analysed by radiologic investigations and clinical progress

IPD SHARING:
Plan to Share IPD: No